CLINICAL TRIAL: NCT05161247
Title: Assessment of the IVF Outcome Parameters After Sperm Selection by Adhesion to Zona Pellucida Proteins
Brief Title: Reproductive Outcome After Sperm Selection for Intracytoplasmic Sperm Injection (ICSI) Using Zona Pellucida Proteins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nadezhda Women's Health Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 59/03122021
Record Dates: First submitted 2021-12-06; First posted 2021-12-17 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Infertility, Male
Keywords: zona pellucida; sperm selection; ICSI; ART outcomes
MeSH Terms: conditions — Infertility, Male | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Intervention Model Description: After couples are recruited for the study they will be randomly allocated to zona selection group (study group) and normal ICSI (control group). For the study group zonae pellucidae from germinal vesicle (GV) or metaphase I (MI) stage oocytes from the female partners will be collected and acid-solubilised to obtain zona proteins. The acid-solubilised zonae will be coated on petri dishes. On the day of their follicular punction the spermatozoa for ICSI in the study group will be selected according to their ability to adhere to the coated zona pellucida proteins from their partner. On the day of their follicular punction the spermatozoa for ICSI in the control group will be selected with no intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zona pellucida sperm selection (Experimental): Semen processing: liquefaction followed by centrifugation and swim-up.
  Zona pellucida sperm selection: Spermatozoa are selected according to their ability to adhere to zona pellucida proteins obtained from their partners native zona pellucida.
  Intracytoplasmic sperm injection (ICSI): Each oocyte is injected with a single morphologically normal spermatozoa. The injection procedure is carried out in a sterilized dish using holding pipette and injection needle.
  Interventions: Other: Zona pellucida sperm selection; Other: Intracytoplasmic Sperm Injection (ICSI)
- Conventional sperm selection (Active Comparator): Semen processing: liquefaction followed by centrifugation and swim-up. Samples are incubated until time of injection.
  Conventional sperm selection: Spermatozoa are selected according to their morphology.
  Intracytoplasmic sperm injection (ICSI): Each oocyte is injected with a single morphologically normal spermatozoa. The injection procedure is carried out in a sterilized dish using holding pipette and injection needle.
  Interventions: Other: Conventional sperm selection; Other: Intracytoplasmic Sperm Injection (ICSI)

INTERVENTIONS:
Other: Zona pellucida sperm selection — Sperm selection for ICSI based on the spermatozoa ability to adhere to immobilized zona pellucida proteins.
  Arms: Zona pellucida sperm selection
Other: Conventional sperm selection — Sperm selection for ICSI based on the sperm morphology.
  Arms: Conventional sperm selection
Other: Intracytoplasmic Sperm Injection (ICSI) — Normal ICSI procedure.

SUMMARY:
The aim of this study is to analyze the effect of a sperm selection method by adhesion to partners' zona pellucida proteins on the assisted reproduction treatment (ART) outcome parameters.

DETAILED DESCRIPTION:
The success rate after treatment by in-vitro fertilisation (IVF) depends on the sperm selection process. Classical sperm selection techniques are based on the spermatozoa morphology and motility, therefore are not able to measure the sperm ability to recognise the oocyte. Furthermore it is known that semen samples showing higher adherence rate to zona pellucida have higher fertilisation potential than spermatozoa that fail to bind to zona proteins.

There have been numerous reports on applying partner' native zona pellucida in sperm selection prior ICSI. However, these studies imply the whole native zona pellucida, while this study will focus on the application of acid-solubilized zonae pellucidae.

Here in this study, the aim is to assess the fertilisation rate, the number and quality of the formed embryos, implantation and ongoing pregnancy success after sperm selection for ICSI by their ability to adhere to immobilized zona pellucida proteins.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis for primary or secondary infertility
* Healthy females
* Clinical diagnosis for unexplained infertility
* Females between 20 and 45 years old.
* Males between 20 and 50 years old.
* At least 3 retrieved oocytes per follicular puncture with at least 1 oocyte at germinal vesicle (GV) or metaphase I (MI) stage

Exclusion Criteria:

* Presence of low quality oocytes
* Females with endometrial or ovarian infertility factor

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 368 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Fertilisation rate | 24 hours after ICSI
  Defined as number of fertilized oocytes (presence of 2 pronuclei) per total number of injected oocytes.
Embryo quality | 2 to 6 days after ICSI
  Morphological evaluation of the cultured embryos will be conducted 120 or 144 hr following sperm injection. Blastocysts scoring will be performed on day 5 or 6 depending on the blastocoel cavity expansion and on the inner cell mass and trophectoderm cells integrity.
Implantation rate | 14 days after embryo transfer
  Defined as high levels of human chorionic gonadotropin (hCG) in the peripheral blood per transfer.
Clinical pregnancy rate | 6 weeks after embryo transfer
  Defined as number of gestational sacs with fetal heart beat, shown by ultrasound in gestational week 6 per number of embryo transferred.

CONTACTS AND LOCATIONS:
Locations (1):
- Nadezhda Women's Health Hospital, Sofia, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No